CLINICAL TRIAL: NCT03975881
Title: Multicenter Open Pilot Study for the Use Smartphone Application to Prevent Suicidal Relapse Among 15-35 Years-old With Previous Suicide Attempted
Brief Title: Study for the Use Smartphone Application to Prevent Suicidal Relapse Among 15-35 Years-old With Previous Suicide Attempted
Acronym: MED COMPANION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Angers (Other Government); Rennes University Hospital (Other); Saint Antoine University Hospital (Other); Université de Nantes (Other); Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC18_0038
Record Dates: First submitted 2018-04-09; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Suicide Attempt by Scalding
Keywords: Suicide attempts; digital device; adolescent; adults
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: Patients aged 15 to 35 who made a suicide attempt and went through the emergency departments of the participating hospitals (Nantes, Angers, Rennes and Poitiers).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): Patients aged 15 to 35 who made a suicide attempt and went through the emergency departments of the participating hospitals (Nantes, Angers, Rennes and Poitiers).
  Interventions: Other: application on smartphone

INTERVENTIONS:
Other: application on smartphone — The aim of this study is to test the feasibility of our approach of preventing suicide relapse with the use of a smartphone application.
  Other Names: MEDICAL COMPANION

SUMMARY:
Context: Suicide is the 2nd cause of death during adolescence Compliance with post SA care is low and variable with effective compliance ranging from 17.5% to 47% . Therefore, prevention programs should also focus on high-risk individuals with a previous history of SA.

Adolescents and young adults are considered to be digital natives, they are therefore a relevant population for the testing of Smartphone Application.

Project: The Investigators propose an innovative and new approach to prevent SA and Suicide for patients, based on a mobile healthcare application.

The program is an add-on to the usual care process.

Study: In a multicentric randomized pilot study with 15 to 35 years-old patients having previous SA, the primary goal for pilot study is to observe the filling rate of the application (feasibility).

DETAILED DESCRIPTION:
Suicide is the 2nd cause of death during adolescence in Europe (1.200/year, 7.9 % of deaths in this age group) and the prevalence of Lifetime Suicide Attempts (SA) in this population is 4.2%. Within a year of the SA, the repetition rate in adolescent populations ranges from 15% to 28%.

Post-SA management is crucial and treatment compliance is a major concern in adolescent populations. A French consensus psychiatric workgroup recommends that when patient is discharged from emergency room (ER) or hospitalization, it is important to organize health care. Unfortunately, these recommendations are imprecise and, moreover, from 40 to 77% of adolescents with previous SAs do not follow the recommendations of the post crisis program. In real clinical practice, patients barely follow the recommended treatment.

Reducing the SA repetition rate and increasing compliance with the recommended post-crisis program are two synergic issues.

The incredible and recent adoption of smartphone health applications (apps), that collect data (weight, exercises…) and allow the consumer to see graphs and diagrams, illustrates the sociological and psychological power of digital self-care and self-management. This phenomenon is particularly important for adolescents and young adults, who are considered to be digital natives. Medical experience is mainly based on the idea that is could be very useful to ask the patient to fill in scales or questionnaires on his/her smartphone instead of on a computer or a paper sheet. This is called Ecological Momentary Assessment (EMA) as it is a naturalistic method to access clinical data.

There are a few positive experiments in self-management (or self-care) using smartphone applications in psychiatry. In the field of suicide and mood disorders they have very interesting and promising results (high filling rates and better compliance to heath care programs). However, despite a few self-care aspects most of these apps are based on psycho-education programs and suffer in reality from lack of feedback.

Second field of apps use is Ecological Momentary intervention (EMI). Main idea is to use EMA data in algorithm in order to produce personalized comments and advises for patients. With the development of machine learning, it is obvious that EMI will have great implication in the future. There are few experiences with EMI but recent reviews all suggest that it is results are promising in mood disorders and anxiety.

The investigators are proposing an EMA + EMI new approach to prevent patient SA and Suicide based on a mobile healthcare application. This application is not connected. This is noticeably different then connected approach, using connected technology (phone, visual-phone and text messages) such as the Suicide Intervention Assisted by Message (SIAM) program, with text messages sent (sometimes automatically) by healthcare professionals to high-risk suicide subjects has shown positive preliminary results, with a reduced repetition rate. The App will be customised for each user when redeemed with a personal code provided by the practitioner. The App will collect data from the patient regarding anxiety, mood and sleep disorders twice a day (with a decreased frequence along the period of use), essentially based on analogic visual scales and drop-down lists. An algorithm-based feedback will pro-actively inform the patient with comments and advice based on WHO recommendations and/or associated with self-coping or Mindfulness practices. The aim is to position the smartphone application like a health care partner, it's name will be Medical Companion.

In order to assess the efficiency of the complete app the investigators will first lead a multicentre open pilot study with 6 months of follow-up in an adolescents and young adults population with a history of suicide attempts.

The application is an association of a "conventional" EMA program and an innovative algorithm-based response to the patient. Built on the notion of self-care, this app is not connected and the patient's responses are processed in the algorithm: (i) to provide feed-back regarding their mental state (contextualized, i.e. "you seem to be less anxious then yesterday") and, (ii) to advice them about what to do (for example "call a friend" "breath deeply 5 times in a row"…). Each mental status will be analysed by the Bayesian application algorithm. Regular evaluations are also provided on screen with easy to see graphs that might be viewed by the patient. These graphs could (and should) be seen by the psychiatrist, or psychologist involved in the Care as Usual program that all participants will still have. In sum, medical practitioners involved in the patient's usual care will have access to synthetic presentation of patient's responses and the investigators plan to ask participants about their experience.

ELIGIBILITY:
Inclusion Criteria:

* Boy or girl, aged 15 to 35 years and having made a suicide attempt within 96 hours requiring emergency admission.
* Informed and signed consent of patient and parents (if applicable)
* Patient affiliated to social security

Exclusion Criteria:

* Patient with a severe psychiatric condition such as, schizophrenia, autistic spectrum disorder and antecedent of more than one suicide attempt (not counting this).
* Patient without smartphone under iOS (mobile operating system developed by Apple) or Android, or without easy access (eg boarding school, social center ...)
* Patient with an intellectual disability making it impossible to use the application (clinically estimated).
* Absence of motivation in relation to the study.
* Patient who does not want or can not give informed consent or understand it.
* Patient whose follow-up seems difficult for psychological, geographical or social reasons, according to the judgment of the investigator
* Not affiliated to social security

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the usage rate of the Medical Companion application over a period of 6 months. | 6 months
  Ratio calculation (r) : r = (number of uses done) / (number of uses expected)

SECONDARY OUTCOMES:
Evaluation of the use rate of the application over 6 months | 6 months
  Frequency of use of the application, data generated automatically by the internal program of the application Medical Companion
Evaluation of the use rate of the application over 6 months | 6 months
  duration of use of the application
Evaluation of suicidal ideation after 6 months of use of the application, | 6 months
  Rate of suicidal ideation at 6 months assessed by telephone call in families using ( 1 to 7)
Evaluation of suicidal recidivism at 6 months | 6 months
  Rate of suicidal recidivism at 6 months evaluated by phone call in families
Assessment of the compliance rate at recommended care | 6 months
  Rate of compliance to recommended care at discharge from hospital (number of appointments honored)
Assessment of the compliance rate at recommended care | 6 months
  Rate of compliance to recommended care at 6 months evaluated by phone call in families
Evaluation of the evolution of the level of sadness of the subject during the 6 months of follow-up | 6 months
  Visual Analogic scale (1 is bad to 10 is perfect ) generated automatically from the subject's responses by the application's internal program
Evaluation of the evolution of the level of sleep disorders of the subject during the 6 months of follow-up | 6 months
  Visual Analogic scale (1 is bad to 10 is perfect ) generated automatically from the subject's responses by the application's internal program.

CONTACTS AND LOCATIONS:
Overall Officials: Fanny GOLLIER BRIANT, Study Chair — Nantes University Hospital
Locations (3):
- France (3):
  - CHU d'Angers, Angers
  - CH Poitiers, Poitiers
  - CH Rennes, Rennes

REFERENCES:
- [Derived] Mouchabac S, Leray P, Adrien V, Gollier-Briant F, Bonnot O. Prevention of Suicidal Relapses in Adolescents With a Smartphone Application: Bayesian Network Analysis of a Preclinical Trial Using In Silico Patient Simulations. J Med Internet Res. 2021 Sep 30;23(9):e24560. doi: 10.2196/24560. PMID 34591030